CLINICAL TRIAL: NCT00328523
Title: Ezetimibe Together With Any Statin Cholesterol Enhancement
Brief Title: TWICE (Ezetimibe Together With Any Statin Cholesterol Enhancement)(0653-060)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653-060; 2006_024
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolaemia; Hyperlipidaemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Ezetimibe; Duration of Therapy

INTERVENTIONS:
Drug: MK-0653, ezetimibe
Drug: Duration of Treatment: 3 months

SUMMARY:
In patients with primary hypercholesterolemia treated with a statin and with ldl-c above the recommended target goal (esc 2003 recommendations ldl>=1.15 g/l) to compare the efficacy and the safety of ezetrol added to ongoing statin and non drug therapeutic intervention (patient motivation on diet or physical activities or both).

ELIGIBILITY:
Inclusion Criteria:

* Primary hypercholesterolemia treated with any statin at any dose, for at least 3 months with a ldl cholesterol above 115 mg/dl (esc 2003 recommendations).

Exclusion Criteria:

* pregnant or breast feeding women
* Lipid-lowering agents including hmg-coa reductase inhibitors other than the current statin, fish oils, cholestyramin, niacin (>200 mg/day) and fibrates taken within the 3 months preceding visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1496 (Actual)
Dates: Start 2004-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Percent of patients attaining the ldl cholesterol target goal based on the lipids result at the end of the study (3 months).

SECONDARY OUTCOMES:
Treatment with ezetimibe 10 mg/day will be well tolerated and no difference in tolerance will be shown between the 3 treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Steg PG, Verdier JC, Carre F, Darne B, Ducardonnet A, Jullien G, Farnier M, Giral P, Haiat R; TWICE Investigators, France. A randomised trial of three counselling strategies for lifestyle changes in patients with hypercholesterolemia treated with ezetimibe on top of statin therapy (TWICE). Arch Cardiovasc Dis. 2008 Nov-Dec;101(11-12):723-35. doi: 10.1016/j.acvd.2008.10.008. Epub 2008 Nov 20. PMID 19059567